CLINICAL TRIAL: NCT02253979
Title: Comparison of VivaSightTM Double Lumen Tube With a Conventional Double Lumen Tube in Adult Patients Undergoing Video Assisted Thoracoscopic Surgery
Brief Title: Comparison of VivaSightTM Double Lumen Tube With a Conventional Double Lumen Tube
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0334-12-RMB_CTIL
Record Dates: First submitted 2014-09-28; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Endotracheal Intubation; Airway Management; One Lung Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard double lumen tube (Placebo Comparator): Intervention: Standard double lumen tube
  Interventions: Device: Standard double lumen tube
- VivaSight double lumen tube (Experimental): Intervention: VivaSight double lumen tube
  Interventions: Device: VivaSight double lumen tube

INTERVENTIONS:
Device: Standard double lumen tube — Endotracheal left side double lumen tube
  Arms: standard double lumen tube
Device: VivaSight double lumen tube — VivaSight double lumen endotracheal intubation
  Arms: VivaSight double lumen tube

SUMMARY:
Double lumen tube (DLT) is an enotracheal tube that facilitates one lung ventilation. The DLT exact position in the airways is verified by fiber-optic bronchoscopy (FOB) after intubation. The VivaSight TM DL is a single use left DLT with a camera embedded in the tube's right side port. This study was designed to compare the VivaSightTM DL to the standard DLT.

DETAILED DESCRIPTION:
Double lumen tube (DLT) is an enotracheal tube that facilitates one lung ventilation. The efficiency of the DLT depends on its exact position in the airways, as verified by fiber-optic bronchoscopy (FOB) after intubation, and re-verified after positioning the patient on the lateral position. The VivaSight TM DL is a single use left DLT with a camera embedded in the tube's right side port. The view from the camera appears continuously on a monitor. This study was designed to compare the VivaSightTM DL to the standard DLT. The primary end point is the time required for intubation with visual confirmation of DLT position.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing video assisted thoracoscopic lung lobectomy

Exclusion Criteria:

* anticipated difficult intubation, patients who required rapid sequence induction
* patients with known tracheal pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Time required for endotracheal intubation with visual confirmation of double lumen tube position position. | During induction of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Dan Levy-Faber, Dr., Principal Investigator — Senior Surgeon, Department of Cardio-Thoracic Surgery

REFERENCES:
- [Result] Heir JS, Purugganan R, Jackson TA, Norman PH, Cata JP, Kosturakis A, Thakar D. A retrospective evaluation of the use of video-capable double-lumen endotracheal tubes in thoracic surgery. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):870-2. doi: 10.1053/j.jvca.2013.11.011. Epub 2014 Mar 20. PMID 24656617
- [Result] Inoue S, Nishimine N, Kitaguchi K, Furuya H, Taniguchi S. Double lumen tube location predicts tube malposition and hypoxaemia during one lung ventilation. Br J Anaesth. 2004 Feb;92(2):195-201. doi: 10.1093/bja/aeh055. PMID 14722168
- [Result] Klein U, Karzai W, Bloos F, Wohlfarth M, Gottschall R, Fritz H, Gugel M, Seifert A. Role of fiberoptic bronchoscopy in conjunction with the use of double-lumen tubes for thoracic anesthesia: a prospective study. Anesthesiology. 1998 Feb;88(2):346-50. doi: 10.1097/00000542-199802000-00012. PMID 9477054